CLINICAL TRIAL: NCT00104403
Title: A Phase II Multicenter, Randomized, Double-blind, Placebo-controlled, Dose-ranging, Parallel Group Study of the Safety and Efficacy of the Oral NeuroKinin-1 Receptor Antagonist, GW679769 in Combination With Ondansetron Hydrochloride and Dexamethasone for the Prevention of Chemotherapy-Induced Nausea
Brief Title: Study Of Prevention of Chemo-Induced Nausea and Vomiting Caused By Moderately Emetogenic Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NKV101983
Record Dates: First submitted 2005-02-28; First posted 2005-03-01 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Nausea and Vomiting, Chemotherapy-Induced; Chemotherapy-Induced Nausea and Vomiting
Keywords: Vomiting; CINV; Emesis; Nausea; Chemotherapy-Induced Nausea and Vomiting
MeSH Terms: conditions — Nausea; Vomiting | interventions — casopitant; Dexamethasone; Ondansetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GW679769
Drug: Dexamethasone
Drug: Ondansetron Hydrochloride
  Other Names: GW679769; Dexamethasone

SUMMARY:
This study was designed to assess the safety and efficacy of different dosages and administration schedules of an investigational agent administered over 3 days when added to standard therapy used in the prevention of chemotherapy-induced nausea and vomiting in cancer patients. Subjects will be asked to complete daily diaries while on study medication. In addition subjects will be required to return to the investigational site several times during the course of the study for follow up safety assessments which may include blood samples for hematology and chemistry evaluations as well as physical exams. A final assessment will be preformed on study Day 20-30 at which time the subject will complete the study.

DETAILED DESCRIPTION:
A Phase II Multicenter, Randomized, Double-blind, Placebo-controlled, Dose-ranging, Parallel Group Study of the Safety and Efficacy of the Oral NeuroKinin-1 Receptor Antagonist, GW679769 in Combination with Ondansetron Hydrochloride and Dexamethasone for the Prevention of Chemotherapy-Induced Nausea and Vomiting in Cancer Subjects Receiving Moderately Emetogenic Chemotherapy

ELIGIBILITY:
Inclusion criteria:

* Willing to provide a written informed consent prior to receiving any study-specific procedures or assessments.
* Diagnosed with a solid malignant tumor and has not previously received chemotherapy.
* Scheduled to receive chemotherapy conducive to regimens outlined in the study protocol.

Exclusion criteria:

* Not received any investigational product within 30 days of enrollment into the study.
* Must not be pregnant.
* Must not be of childbearing potential or is willing to use specific barrier methods outlined in the protocol.
* Must not be scheduled to receive radiation therapy to the abdomen or to the pelvis within seven (7) days prior to starting study medication.
* Must not be currently under treatment for a condition which may cause nausea or vomiting (i.e., active peptic ulcer disease, gastric obstruction).
* Must not have a history of peptic ulcer disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 722 (Actual)
Dates: Start 2004-12; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Based on the number of subjects who do not experience vomiting, retching or nausea over a 5 day period following the initiation of chemotherapy.

SECONDARY OUTCOMES:
Based on routine physical exam findings, vital signs, routine clinical laboratory tests, clinical monitoring and/or observation, and adverse events reporting performed during scheduled visits.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (101):
- United States (46):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Corona, California
  - GSK Investigational Site, Greenbrae, California
  - GSK Investigational Site, Loma Linda, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Palm Springs, California
  - GSK Investigational Site, Lakewood, Colorado
  - GSK Investigational Site, Boynton Beach, Florida
  - GSK Investigational Site, Hudson, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Ocala, Florida
  - GSK Investigational Site, Centralia, Illinois
  - GSK Investigational Site, Park Ridge, Illinois
  - GSK Investigational Site, Skokie, Illinois
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, Muncie, Indiana
  - GSK Investigational Site, New Albany, Indiana
  - GSK Investigational Site, Hutchinson, Kansas
  - GSK Investigational Site, Alexandria, Louisiana
  - GSK Investigational Site, Baton Rouge, Louisiana
  - GSK Investigational Site, Bethesda, Maryland
  - GSK Investigational Site, Worcester, Massachusetts
  - GSK Investigational Site, Bay City, Michigan
  - GSK Investigational Site, Tupelo, Mississippi
  - GSK Investigational Site, Jefferson City, Missouri
  - GSK Investigational Site, Rolla, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Sparta, New Jersey
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Bismarck, North Dakota
  - GSK Investigational Site, Akron, Ohio
  - GSK Investigational Site, Canton, Ohio
  - GSK Investigational Site, Sumter, South Carolina
  - GSK Investigational Site, Corpus Christi, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Tyler, Texas
  - GSK Investigational Site, Ogden, Utah
  - GSK Investigational Site, West Point, Utah
  - GSK Investigational Site, Burlington, Vermont
  - GSK Investigational Site, Abingdon, Virginia
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Everett, Washington
  - GSK Investigational Site, Tacoma, Washington
  - GSK Investigational Site, Rhinelander, Wisconsin
- Argentina (2):
  - GSK Investigational Site, Capital Federal, Buenos Aires
  - GSK Investigational Site, Buenos Aires
- Austria (2):
  - GSK Investigational Site, Salzburg
  - GSK Investigational Site, Vienna
- Canada (5):
  - GSK Investigational Site, Kitchener, Ontario
  - GSK Investigational Site, Oshawa, Ontario
  - GSK Investigational Site, Charlottetown, Prince Edward Island
  - GSK Investigational Site, Greenfield Park, Quebec
  - GSK Investigational Site, Québec, Quebec
- GSK Investigational Site, Santiago, Región Metro de Santiago, Chile
- GSK Investigational Site, Osijek, Croatia
- Czechia (3):
  - GSK Investigational Site, Hradec Králové
  - GSK Investigational Site, Ostrava - Poruba
  - GSK Investigational Site, Prague
- Germany (3):
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Regensburg, Bavaria
  - GSK Investigational Site, Essen, North Rhine-Westphalia
- Greece (3):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Haidari
  - GSK Investigational Site, Thessaloniki
- GSK Investigational Site, Pokfulam, Hong Kong
- Hungary (2):
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Mátraháza
- Ireland (3):
  - GSK Investigational Site, Dublin
  - GSK Investigational Site, Tallaght, Dublin
  - GSK Investigational Site, Tullamore
- Mexico (2):
  - GSK Investigational Site, Durango, Durango
  - GSK Investigational Site, Mérida, Yucatán
- Pakistan (2):
  - GSK Investigational Site, Karachi
  - GSK Investigational Site, Lahore
- Philippines (2):
  - GSK Investigational Site, Quezon City
  - GSK Investigational Site, Taft Avenue, Manila
- Poland (4):
  - GSK Investigational Site, Kielce
  - GSK Investigational Site, Olsztyn
  - GSK Investigational Site, Opole
  - GSK Investigational Site, Szczecin
- GSK Investigational Site, Lisbon, Portugal
- Russia (2):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Moscow Region
- GSK Investigational Site, Singapore, Singapore
- Slovakia (2):
  - GSK Investigational Site, Bratislava
  - GSK Investigational Site, Žilina
- Spain (4):
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Marid
  - GSK Investigational Site, Pontevedra
  - GSK Investigational Site, Valencia
- Taiwan (2):
  - GSK Investigational Site, Tainan
  - GSK Investigational Site, Taipei
- Thailand (2):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Chiang Mai
- United Kingdom (5):
  - GSK Investigational Site, Exeter, Devon
  - GSK Investigational Site, Chelmsford, Essex
  - GSK Investigational Site, Cardiff, Glamorgan
  - GSK Investigational Site, Edinburgh, Midlothian
  - GSK Investigational Site, Shrewsbury

REFERENCES:
- [Result] Arpornwirat W, Albert I, Hansen VL, Levin J, Bandekar RR, Grunberg SM. Phase 2 trial results with the novel neurokinin-1 receptor antagonist casopitant in combination with ondansetron and dexamethasone for the prevention of chemotherapy-induced nausea and vomiting in cancer patients receiving moderately emetogenic chemotherapy. Cancer. 2009 Dec 15;115(24):5807-16. doi: 10.1002/cncr.24630. PMID 19834961